CLINICAL TRIAL: NCT04617392
Title: Research of Sarcopenia in Patients After Bariatric-metabolic Surgery - the Effect of Programmed Aerobic and Power Exercising on the Functionality, Volume and Morphology of Muscle Tissue
Brief Title: Bariatric-metabolic Surgery - the Effect of Postoperative Exercising on Sarcopenia
Acronym: SarxOb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Masaryk University (Other)
Collaborators: Hospital AGEL Ostrava-Vitkovice (Unknown); University of Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SarxOb_2020
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Sarcopenia; Obesity; Sarcopenic Obesity
Keywords: obesity; bariatric surgery; weight loss; sarcopenia; muscle; exercise; magnetic resonance imaging; gait; kinematics; kinetics; cartilage surfaces
MeSH Terms: conditions — Sarcopenia; Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlled group (Active Comparator): 25 patients after bariatric-metabolic surgery without controlled postprocedural training
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- active group (Experimental): 25 patients after bariatric-metabolic surgery with controlled postprocedural training
  Interventions: Procedure: Laparoscopic sleeve gastrectomy; Other: Strength endurance training

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Sleeve gastrectomy involves removing a part of the stomach, limiting the amount of food the patient can eat.
Other: Strength endurance training — Patients included in the active cohort arm with physical activity will undergo three months of strength endurance training under the supervision of a professional physiotherapist
  Arms: active group

SUMMARY:
The investigators' study published in 2020 (Pekar, M. et al.: The risk of sarcopenia 24 months after bariatric surgery - assessment by dual energy X-ray absorptiometry (DEXA): a prospective study; Videosurgery Miniinv 2020; https://doi.org/10.5114/wiitm.2020.93463) shows that patients are at risk of sar-copenia after bariatric-metabolic (BM) surgery. BM surgery leads to significant changes in body composition. Significant fat loss is followed by unwanted muscle loss. The study shows that the lack of physical activity is typical for these patients. To the algorithm of postoperative care the investigators plan to include controlled exercise programs for these patients. The investigators do not know what the complexity and time required to keep patients in good condition and reduce the risk of sarcopenia is. The investigators want to find the adequate amount of physical activity while maintaining long-term compliance of these patients.

DETAILED DESCRIPTION:
Obesity is an important medical problem. The number of obese individuals is increasing continuously in response to various environmental and genetic factors. For some morbidly obese patients, surgery is the only effective type of therapy. Despite bariatric surgery having good outcomes in terms of weight loss, it is associated with some adverse effects: several studies have reported subsequent alterations in bone and muscle metabolism, patients are getting in risk of sarcopenia. Of the surgical techniques available (laparoscopic gastric banding, Roux-en-Y bypass, biliopancreatic diversion), laparoscopic sleeve gastrectomy (LSG) is currently the technique of choice. This type of surgery leads to significant changes in body composition. Significant fat loss is followed by unwanted muscle loss. To the algorithm of postoperative care the investigators plan to include controlled exercise programs for these patients. The investigators do not know what the complexity and time required to keep patients in good condition and reduce the risk of sarcopenia is. The investigators want to find the adequate amount of physical activity while maintaining long-term compliance of these patients.

The study has been designed as a prospective randomized study, which is in conformity with the principles and guidelines of the Helsinki Declaration, good clinical practice and will be approved by the Ethical Committee of the Hospital AGEL Ostrava-Vitkovice, Czech Republic.

Potential study participants will undergo an initial examination at the clinical department of the surgical department specializing in obesity. In addition to professional surgical and internal examination, the potential patient will be examined by a clinical psychologist for the ability to participate in this type of study for a long time. Informed consent will be provided to selected study participants.

50 patients who undergo surgery will be randomized in two cohorts:

* Cohort 1: obese patients with LSG: 25 patients with controlled aerobic / anaerobic activity
* Cohort 2: obese LSG patients 25 patients without controlled physical activity

The patients enrolled in the study are followed for the period of 24 months. Individual will be evaluated before the bariatric procedure and 3, 6, 12, 18 and 24 months after the procedure.

Primary goal of the study is to evaluate the Hypothesis 0 : there is no difference between muscle function, volume and morphology between patients after BM operations who are no longer controlled by physical activity and between patients who undergo controlled regular exercise programs under professional supervision.

Secondary objectives: Monitoring of knee cartilage during weight reduction after bariatric surgery and monitoring of gait biomechanics during weight reduction after bariatric surgery

Patients undergo the following examinations:

Weight: body weight will be measured on a calibrated scale. The measurement itself will be performed in underwear, without shoes.

Waist circumference: the circumference will be measured using a fixed tape measure.

Body composition: measurement of body composition of obese individuals will be performed using DXA (Dual-emission X-ray absorptiometry, Discovery A, Hologic).

Examination of muscle mass and muscle strength:

* Muscle mass: measurement of the composition and structure of skeletal muscles and fat in the thigh will be performed using MRI (Magnetic Resonance Imaging)
* Muscle strength: the measurement will be performed using a battery of tests:

handgrip dynamometer, chair-stand-walk test, test of getting up from a chair, test of 400 meters walk

Physical activity:

* physical activity questionnaire
* controlled regular exercise programs: patients will be divided into two cohorts - with and without physical intervention. Patients included in the intervention cohort with physical activity will undergo three months of strength endurance training under the supervision of a professional physiotherapist.

Quality of life: calibrated 36-Item Short Form Health Survey (SF-36) and The Impact of Weight on Quality of Life (IWQOL) questionnaire

Biochemical analyzes:

Blood samples will be taken from each test subject after 12 hours of fasting by venipuncture before the actual bariatric procedure and then repeatedly in the follow-up period after the procedure. The samples will be centrifuged under standard conditions and the concentrations of the following substances will then be determined in the serum samples:

• glucose, glycated hemoglobin, alkaline phosphatase, total calcium, phosphates, parathyroid hormone, total protein, albumin, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyltransferase, creatinine. After determination of these analytes, serum (plasma) aliquots will be frozen at -80 ° C until analysis of other selected parameters.

WITHDRAWAL FROM THE STUDY

Persons involved in the study may terminate their participation or be excluded from the study at any time for the following reasons:

* Death of the subject
* Voluntary withdrawal from the study: the subject voluntarily decides not to continue in the next part of the study.
* Loss from follow-up: the subject does not show up for scheduled inspections more than one month after the scheduled inspection or examination.
* Risk / benefit ratio: while evaluating the results during follow-up, the clinical coordinator finds that continuing the study is not in the best interests of the subject with respect to the subject.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 30-50 kg/m2
* ability to understand informed consent
* signed informed consent
* patient's residence within 100 km from Ostrava Czech Republic

Exclusion Criteria:

* History of gastric surgery
* acute gastric ulcers or inflammation
* Type 1 Diabetes mellitus
* celiac disease
* history of malignity
* previous bariatric-metabolic surgery or endoscopic obesity treatment,
* specific genetic and humoral diseases connected to obesity (Prader-Willi syndrome, mutation of melanocortin receptor 4, etc.)
* history of knee surgery
* non MRI compatible patients' devices and implants
* severe hematological diseases
* acute or chronic pancreatitis
* cirrhosis
* severe psychiatric diseases
* uncontrolled hypertense
* immunological diseases
* long-term corticoid therapy
* uncontrolled thyroid diseases
* renal insufficiency
* alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of lean mass by DXA measures (in kg/m2) | 24 months
  higher values mean better result
fat infiltration of muscles by MRI (in %) | 24 months
  lower content of fat means better result
muscle strength by handgrip dynamometer (in kg) | 24 months
  higher values in this physical performance test mean better result
muscle strength by walk test (in m) | 24 months
  higher values in this physical performance test mean better result
muscle strength by Timed Up and Go test (in s) | 24 months
  lower values in this physical performance test mean better result
thickness of cartilage surface of the knee by MRI (in mm) | 24 months
  higher values mean better result

SECONDARY OUTCOMES:
changes of fat mass by DXA measures (in kg/m2) | 24 months
  lower values mean better result

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaudart C, Dawson A, Shaw SC, Harvey NC, Kanis JA, Binkley N, Reginster JY, Chapurlat R, Chan DC, Bruyere O, Rizzoli R, Cooper C, Dennison EM; IOF-ESCEO Sarcopenia Working Group. Nutrition and physical activity in the prevention and treatment of sarcopenia: systematic review. Osteoporos Int. 2017 Jun;28(6):1817-1833. doi: 10.1007/s00198-017-3980-9. Epub 2017 Mar 1. PMID 28251287
- [Background] Bosaeus I, Rothenberg E. Nutrition and physical activity for the prevention and treatment of age-related sarcopenia. Proc Nutr Soc. 2016 May;75(2):174-80. doi: 10.1017/S002966511500422X. Epub 2015 Dec 1. PMID 26620911
- [Background] CARSOTE, Mara, Razvan PETRESCU, Adriana Elena NICA, Adina GHEMIGIAN, Dan Nicolae PADURARU a Ana VALEA. BARIATRIC SURGERY AND OSTEOPO-ROSIS. Romanian Medical Journal [online]. 2016, 63(4), 297-299 [cit. 2020-10-12]. ISSN 12205478.
- [Background] CARVALHO, Nara, Vinícius BACCIN, Narriane HOLANDA, João FILHO, Marta CA-RVALHO, Gitana SILVA, Flávia PIMENTA a José ALVES. SUN-542 Comparison of Different Muscle Mass Indices for Evaluation of Low Muscle Mass Regarding Muscle Function, Bone Mineral Density and Metabolic Profile in Obese Patients Prior to Bariatric Surgery. Journal of the Endocrine Society [online]. 2019, 3 [cit. 2020-10-12]. ISSN 24721972.
- [Background] CARVALHO, Nara, Caio LIMEIRA, Vinícius BACCIN, et al. SAT-LB018 Different Definitions of Sarcopenia and Its Correlations with Anthropometric Measure-ments, Body Composition, Handgrip Strength, Metabolic Profile and Bone Mine-ral Density in Obese Women. Journal of the Endocrine Society [online]. 2019, 3
- [Background] Ciudin A, Simo-Servat A, Palmas F, Barahona MJ. Sarcopenic obesity: a new challenge in the clinical practice. Endocrinol Diabetes Nutr (Engl Ed). 2020 Dec;67(10):672-681. doi: 10.1016/j.endinu.2020.03.004. Epub 2020 Jun 18. English, Spanish. PMID 32565081
- [Background] Dantas WS, Roschel H, Murai IH, Gil S, Davuluri G, Axelrod CL, Ghosh S, Newman SS, Zhang H, Shinjo SK, das Neves W, Merege-Filho C, Teodoro WR, Capelozzi VL, Pereira RM, Benatti FB, de Sa-Pinto AL, de Cleva R, Santo MA, Kirwan JP, Gualano B. Exercise-Induced Increases in Insulin Sensitivity After Bariatric Surgery Are Mediated By Muscle Extracellular Matrix Remodeling. Diabetes. 2020 Aug;69(8):1675-1691. doi: 10.2337/db19-1180. Epub 2020 May 14. PMID 32409493
- [Background] Delgado Andre L, Basso-Vanelli RP, Di Thommazo-Luporini L, Angelica Ricci P, Cabiddu R, Pilon Jurgensen S, Ricardo de Oliveira C, Arena R, Borghi-Silva A. Functional and systemic effects of whole body electrical stimulation post bariatric surgery: study protocol for a randomized controlled trial. Trials. 2018 Oct 31;19(1):597. doi: 10.1186/s13063-018-2844-8. PMID 30382930
- [Background] Esposito A, Campana L, Palmisano A, De Cobelli F, Canu T, Santarella F, Colantoni C, Monno A, Vezzoli M, Pezzetti G, Manfredi AA, Rovere-Querini P, Del Maschio A. Magnetic resonance imaging at 7T reveals common events in age-related sarcopenia and in the homeostatic response to muscle sterile injury. PLoS One. 2013;8(3):e59308. doi: 10.1371/journal.pone.0059308. Epub 2013 Mar 12. PMID 23555016
- [Background] Gray C, MacGillivray TJ, Eeley C, Stephens NA, Beggs I, Fearon KC, Greig CA. Magnetic resonance imaging with k-means clustering objectively measures whole muscle volume compartments in sarcopenia/cancer cachexia. Clin Nutr. 2011 Feb;30(1):106-11. doi: 10.1016/j.clnu.2010.07.012. Epub 2010 Aug 19. PMID 20727625
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30312372/